CLINICAL TRIAL: NCT05098665
Title: PATHWAY-RCT: Preventing Admission To Hospital With Attr cardiomyopathY Using Remote Cardiac Telemonitoring
Brief Title: PATHWAY-RCT: Preventing Admission To Hospital With Attr cardiomyopathY
Acronym: PATHWAY-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Richmond Research Institute (Industry)
Collaborators: Richmond Pharmacology Limited (Industry); National Amyloidosis Centre (Unknown)
Responsible Party: Sponsor
Organization: Richmond Pharmacology Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C21026
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial of telemonitoring intervention versus usual care
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask this type of intervention for participant or care provider, but outcomes will be assessed in a blinded fashion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - RCT telemonitoring (Active Comparator): 160 ATTR-CM patients assigned to receive telemonitoring intervention
  Interventions: Combination Product: Telemonitoring service
- Arm B - RCT usual care (No Intervention): Control group of 160 ATTR-CM patients assigned to receive usual care

INTERVENTIONS:
Combination Product: Telemonitoring service — Patients in the active arm will receive a cellular network connected set of digital scales, and instructed to take their weight each morning at the same time. This device (BodyTrace) automatically uploads each daily weight reading to a central database. A clinical algorithm is applied to detect those at risk of acute and subacute decompensated heart failure. Patients are contacted within 24-48 hours of being flagged as at risk by a heart failure specialist. A clinical history is taken, and medication review undertaken, in line with a protocol. Diuretics are adjusted as per the protocolised changes, or for patients at ceiling of treatment, referral for local specialist review is made. A third protocol for follow-up is then followed to close the loop of intervention.
  Arms: Arm A - RCT telemonitoring

SUMMARY:
Cardiac amyloidosis is a condition where the heart muscle, amongst other tissues, is infiltrated by the abnormal build-up of proteins called amyloid. This stiffens and thickens the heart muscle over time which makes it less efficient and puts further stress and strain on the other chambers of the heart, leading to heart failure. The commonest form, that affects predominantly the elderly, is called 'wild-type' ATTR amyloid (TTR is the protein that accumulates). In this condition a patient has a 60% chance of admission to hospital each year after diagnosis. There is no current treatment for ATTR amyloid other than using water tablets to reduce excess fluid and prevent more serious fluid build up in lungs and other tissues. Increasing body weight is the most reliable clinical sign of this fluid build up.

Tele-monitoring is the practice of monitoring patients from a distance and has been shown to reduce heart failure admissions and death in patients with heart failure from any cause. Due to reduced access to primary and secondary care during COVID-19 the investigators instigated tele-monitoring of heart failure in ATTR amyloid patients. This appeared to be an effective intervention in the pilot study. The investigators propose to monitor the weight of patients with cardiac amyloidosis at home and intervene where a build up of fluid is observed by telephone discussion with a doctor. The investigators propose to evidence this in a prospective clinical trial. The investigators will evaluate the effect fairly by comparing tele-monitoring with usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 at the date of signing informed consent which is defined as the beginning of the Screening Period.
2. An established diagnosis of ATTR cardiomyopathy as defined by protocol.
3. Ability to provide written, personally signed and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (R2) (2016) and applicable regulations, before completing any study-related procedures.
4. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
5. Currently a patient at a study site (NAC).

Exclusion Criteria:

1. An inability to have or use BodyTrace device scales at usual residence (for example no mobile network cellular signal)
2. On dialysis or end-stage renal failure (eGFR <25mL/min)
3. Serum albumin <20g/dL or other non-hypervolaemia cause of tissue oedema (e.g. protein-losing enteropathy, nephrotic syndrome)
4. Use of greater than 2 oral diuretics (e.g. on maximum oral diuretic therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Heart-failure related hospitalisations | Study duration (3 years)
  Hospitalisation which can be attributed to heart failure
All-cause mortality | Study duration (3 years)
  Death by any cause, as an annual event rate

SECONDARY OUTCOMES:
All-cause hospitalisation | Study duration (3 years)
  Hospitalisation for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Rezk, MBBS MRCP PhD, Principal Investigator — National Amyloidosis Centre, Royal Free Hospital
Locations (1):
- Richmond Research Institute, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Sharing of personal data with other organisations is not planned